CLINICAL TRIAL: NCT02422823
Title: Comparative Evaluation of the Anesthetic Efficacy of 1,8mL and 3,6mL of 4% Articaine With 1: 100,000 Epinephrine in Blocking the Inferior Alveolar Nerve in Patients With Irreversible Pulpitis of Mandibular Molars
Brief Title: Anesthetic Efficacy of 1,8mL and 3,6mL of Articaine in Inferior Alveolar Nerve Block in Irreversible Pulpitis
Acronym: Volumes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isabel Peixoto Tortamano (Other)
Responsible Party: Sponsor-Investigator, Isabel Peixoto Tortamano, Associate Professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Volumes
Record Dates: First submitted 2015-03-27; First posted 2015-04-21 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-05

CONDITIONS: Pulpitis
Keywords: anesthesia; volumes; articaine; Inferior alveolar nerve block
MeSH Terms: conditions — Pulpitis | interventions — Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- injection of 1.8mL (Experimental): injections of 1.8 mL of 4% articaine with 1:100,000 epinephrine Intervention: inferior alveolar nerve block injection
  Interventions: Drug: Articaine; Drug: Epinephrine
- injection of 3.6mL (Experimental): injections of 3.6 mL of 4% articaine with 1:100,000 epinephrine Intervention: inferior alveolar nerve block injection
  Interventions: Drug: Articaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Articaine — Injection of 1.8mL of 4% articaine with 1: 100,000 epinephrine in block the inferior alveolar nerve in patients with irreversible pulpitis of mandibular molar in 40 patients
  Other Names: Articaine 100, DFL, Rio de Janeiro, RJ, Brasil
  Arms: injection of 1.8mL
Drug: Articaine — Injection of 3.6mL of 4% articaine with 1: 100,000 epinephrine in block the inferior alveolar nerve in patients with irreversible pulpitis of mandibular molar in 40 patients
  Other Names: Articaine 100, DFL, Rio de Janeiro, RJ, Brasil
  Arms: injection of 3.6mL
Drug: Epinephrine

SUMMARY:
Ninety patients with irreversible pulpitis diagnostic will participate in this clinical study. The participants will be divided into 2 groups of 45 patients, who will receive the inferior alveolar nerve block injections of 1.8 mL of 4% articaine (Articaine 100; DFL, Rio de Janeiro, RJ, Brazil) with 1:100,000 epinephrine or 3.6mL of the same solution. Two consecutive negative responses to the maximum pulp stimulus (80 µA) at the electric pulp test were the criterion to determine a pulpal anesthesia as successful. Ten minutes after the IAN block, subjective lip anesthesia will be evaluated by asking the patient whether his/her lip was numb. Thereafter and immediately before the pulpectomy, the electric pulp stimulations will be repeated to determine pulpal anesthesia. During the pulpectomy procedure, the patients were instructed to report any painful discomfort. To evaluate the intensity of pain during the pulpectomy, a verbal analogue scale will be used. The anesthesia will be defined as successful when the dentist accessed the pulp chamber without pain being reported by the patient. In these cases, the pulpectomy will be continued. If report pain will classified the IAN block as unsuccessful.

DETAILED DESCRIPTION:
Ninety patients will Participate in this clinical study. The patients will be admitted to the Emergency Center of the School of Dentistry at the University of São Paulo with a clinical diagnosis of irreversible pulpitis, The study was approved by the Committee on the Ethics of Research on Human Beings of the School of Dentistry at the University of São Paulo (protocol 95/07), and each patient will be informed to sing consent to participate in the study. The 90 participants will be divided into 2 groups of 45 patients, who will receive the inferior alveolar nerve block injections of 1.8 mL (equivalent to 1 cartridge) of 4% articaine (Articaine 100; DFL, Rio de Janeiro, RJ, Brazil) with 1:100,000 epinephrine or 3.6mL (equivalent to 2 cartridges) of the same solution. Two consecutive negative responses to the maximum pulp stimulus (80 µA) at the electric stimulation were the criterion to determine a pulpal anesthesia as successful. Before the IAN block injections, the tooth with irreversible pulpitis, the adjacent tooth, and the contralateral canine will be tested for pulp vitality with an electric pulp test (Vitality Scanner 2006; SybronEndo, Orange, CA). The electric pulp stimulation of the contralateral canine, which will be not anesthetized, will be used as control to ensure that the equipment is working properly and that patients is responding adequately.

The average injection time for each cartridge was approximately 2 minutes. Ten minutes after the IAN block, subjective lip anesthesia will be evaluated by asking the patient whether his/her lip was numb. Thereafter and immediately before the pulpectomy, the electric pulp stimulations will be repeated to determine pulpal anesthesia. During the pulpectomy procedure, the patients were instructed to report any painful discomfort. To evaluate the intensity of pain during the pulpectomy, a verbal analogue scale will be used: 0, no pain; 1, mild, bearable pain; 2, moderate, unbearable pain; 3, severe, intense, and unbearable pain. The anesthesia will be defined as successful when the dentist accessed the pulp chamber without pain being reported by the patient (pain scores 0 or 1). In these cases, the pulpectomy will be continued. Pain scores of 2 or 3 will classified the IAN block as unsuccessful.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-50 years, with mandibular molars with irreversible pulpitis, and have 1 molar adjacent to a molar presenting irreversible pulpites and a healthy contralateral canine with no deep carious lesions, extensive restoration, advanced periodontal disease, a history of trauma, or sensitivity.

Exclusion Criteria:

* Patients who took medication potentially interacting with the anesthetic used in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain measured by a verbal analog scale | intraoperative

SECONDARY OUTCOMES:
Presence of pulpal anesthesia by pulp electrical test | 10 minutes after the block
Patient's report for anesthesia on lip | 10 minutes after the block

CONTACTS AND LOCATIONS:
Overall Officials: Isabel P Tortamano, Principal Investigator — University of Sao Paulo
Locations (1):
- Faculdade de Odontologia da USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Silva SA, Horliana ACRT, Pannuti CM, Braz-Silva PH, Bispo CGC, Buscariolo IA, Rocha RG, Tortamano IP. Comparative evaluation of anesthetic efficacy of 1.8 mL and 3.6 mL of articaine in irreversible pulpitis of the mandibular molar: A randomized clinical trial. PLoS One. 2019 Jul 31;14(7):e0219536. doi: 10.1371/journal.pone.0219536. eCollection 2019. PMID 31365529